CLINICAL TRIAL: NCT00436150
Title: Preventing Postpartum Depression in Adolescent Mothers
Brief Title: Interpersonal Therapy-Based Treatment to Prevent Postpartum Depression in Adolescent Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, maureen phipps, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH077588 (NIH); R34MH077588 (NIH); DSIR 84-CTP
Record Dates: First submitted 2007-02-14; First posted 2007-02-16 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Depression
Keywords: Adolescents; Depression, postpartum
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Participants will receive interpersonal therapy-based treatment
  Interventions: Behavioral: Interpersonal therapy-based treatment
- B (Active Comparator): Participants will receive standard care
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Interpersonal therapy-based treatment — Participants assigned to receive interpersonal therapy-based treatment will focus on the psychological aspects of pregnancy and factors that may play a role in the development of postpartum depression in teenage mothers, such as poor social support, role transitions, and life stressors. Both groups will attend weekly 1-hour sessions for 5 weeks.
  Other Names: REACH
  Arms: A
Behavioral: Standard care — Participants assigned to receive standard care will focus more on the health issues associated with pregnancy and postpartum. Both groups will attend weekly 1-hour sessions for 5 weeks.
  Other Names: Baby Basics
  Arms: B

SUMMARY:
This study will aim to prevent postpartum depression in pregnant teenagers through an interpersonal therapy-based program.

DETAILED DESCRIPTION:
Postpartum depression is believed to be one of the most common complications after pregnancy. This type of depression often occurs within the first year after the baby is born and is most likely caused by dramatic changes in hormone levels after pregnancy. Pregnant teenagers are even more at risk for experiencing complications throughout pregnancy and parenting difficulties after delivery. Minimal research has been done on preventive ways to reduce postpartum depression in teenagers. Therefore, this study will evaluate the effectiveness of an interpersonal therapy-based program at preventing postpartum depression in financially disadvantaged pregnant teenagers.

Participants will first undergo a 15-minute interview about their background and emotions. Participants will undergo a second interview and then be randomly assigned to receive either interpersonal therapy-based treatment or standard care. Participants assigned to receive interpersonal therapy-based treatment will focus on the psychological aspects of pregnancy and factors that may play a role in the development of postpartum depression in teenage mothers, such as poor social support, role transitions, and life stressors. Participants assigned to receive standard care will focus more on the health issues associated with pregnancy and postpartum. Both groups will attend weekly 1-hour sessions for 5 weeks. Homework may be assigned to review topics discussed, and all participants will receive the book Baby Basics. Following treatment, participants will meet with researchers again when they are 34 to 36 weeks pregnant; in the hospital after the baby is born; and 6, 12, and 24 weeks after the baby is born.

ELIGIBILITY:
Inclusion Criteria:

* Less than 24 weeks pregnant
* Not currently being treated for depression
* Speaks and reads English fluently

Exclusion Criteria:

* Currently receiving mental health services from a health care provider
* Meets DSM-IV criteria for an affective disorder, substance use disorder, or psychosis

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Postpartum depression diagnosis | Measured at pretreatment; Weeks 34 to 36 during pregnancy; hospital stay after delivery; and Weeks 6, 12, and 24 postpartum

SECONDARY OUTCOMES:
Degree of depressive symptoms | Measured at pretreatment; Weeks 34 to 36 during pregnancy; hospital stay after delivery; and Weeks 6, 12, and 24 postpartum
Prenatal distress | Measured at pretreatment; Weeks 34 to 36 during pregnancy; hospital stay after delivery; and Weeks 6, 12, and 24 postpartum
Social support | Measured at pretreatment; Weeks 34 to 36 during pregnancy; hospital stay after delivery; and Weeks 6, 12, and 24 postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Phipps, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States